CLINICAL TRIAL: NCT07235033
Title: A Multi-part, Multi-center PLATform Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of Anti-malarial Agents Administered as Monotherapy and/or Combination Therapy IN Participants With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Platform Study to Evaluate the Efficacy and Safety of Anti-malarial Agents in Participants With Uncomplicated Plasmodium Falciparum Malaria (Cohort B2)
Acronym: PLATINUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CADPT13A12201_B2
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: single dose cure malaria; uncomplicated malaria; Plasmodium falciparum; platform study; PLATINUM
MeSH Terms: conditions — Malaria, Falciparum | interventions — NITD 609; Artemether, Lumefantrine Drug Combination; ganaplacide

STUDY DESIGN:
Masking Description: This study is open-label, but Core Clinical Team is blinded to treatment information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort B2: KLU156 + cipargamin (Experimental): Cohort B2: KLU156 + cipargamin
  Interventions: Drug: Cipargamin; Drug: KLU156
- Cohort B2: SoC (Coartem) (Active Comparator): Cohort B2: SoC (Coartem)
  Interventions: Drug: SoC (Coartem)

INTERVENTIONS:
Drug: Cipargamin — oral capsules administered in combination with KLU156
  Other Names: KAE609
  Arms: Cohort B2: KLU156 + cipargamin
Drug: SoC (Coartem) — Standard of Care (Coartem)
  Arms: Cohort B2: SoC (Coartem)
Drug: KLU156 — oral sachet formulation administered in combination with cipargamin
  Other Names: ganaplacide + lumefantrine SDF
  Arms: Cohort B2: KLU156 + cipargamin

SUMMARY:
This is Cohort B2 of the Platform study (NCT05750628) to evaluate the efficacy and safety of Cipargamin + KLU156 in participants with uncomplicated Plasmodium falciparum malaria

DETAILED DESCRIPTION:
The Cohort B2 of this Platfom study (NCT05750628) is the open-label, randomized, two-arm combination therapy evaluating a single oral dose of up to three anti-malarial agents as a loose combination vs. standard of care (SoC), Coartem in adult and adolescent participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥12 years of age at screening.
2. Patients must have acute uncomplicated P. falciparum malaria mono infection at screening confirmed by a parasite count between 1,000 to 150,000 asexual parasite count/μl of blood for P. falciparum.
3. Patients must weigh between 35 kg and 90 kg at screening.
4. Axillary temperature ≥ 37.5ºC or oral/tympanic/rectal temperature ≥ 38.0ºC; or history of fever during the previous 24 hours.

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria at screening or mixed Plasmodium infection (i.e., infection with more than one malaria species) at screening
2. Moderate to severe anemia, chronic hemoglobinopathy (Hemoglobin level < 8 g/dL), or known chronic underlying disease such as sickle cell disease at screening
3. Known clinically significant liver disease (e.g., chronic hepatitis, liver cirrhosis (compensated or decompensated), history of hepatitis B or C, hepatitis A or B vaccination in the last 3 months, known gallbladder or bile duct disease, acute or chronic pancreatitis. Clinical or laboratory evidence of any of the following at screening:

   * AST/ALT > 3 x the upper limit of normal range (ULN), regardless of the level of total bilirubin
   * AST/ALT > 1.5 and ≤ 2 x ULN and total bilirubin is > ULN
   * Total bilirubin > 2 x ULN, regardless of the level of AST/ALT
4. Any known/suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection at screening.
5. Pregnant or nursing (lactating) women, women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using methods of effective contraception, and sexually active patients not willing to practice effective contraception.
6. History or current diagnosis of ECG abnormalities indicating significant risk of safety for patients participating in the study such as:

   * Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker
   * History of familial long QT syndrome or known family history of Torsades de Pointe.
   * Resting heart rate (physical exam or 12 lead ECG) < 50 bpm

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Polymerase chain reaction (PCR) corrected adequate clinical and parasitological response (ACPR) | Day 29
  ACPR is defined as the absence of parasitemia on Study Day 29 irrespective of axillary temperature, without previously meeting any of the criteria of Early Treatment Failure (ETF) or Late Clinical Failure (LCF) or Late Parasitological Failure (LPF).

SECONDARY OUTCOMES:
Parasite clearance time (PCT) | up to Day 7
  To assess the parasite clearance time (PCT) of oral anti malarial agent versus the standard of care (SoC) in participants with uncomplicated P. falciparum malaria
PCR-uncorrected ACPR | Day 29
  To assess the 28-day cure rate of an anti malarial agent administered orally as combination therapy versus the SoC in participants with uncomplicated P. falciparum malaria.
Area under the concentration-time curve from time zero to the last measurable concentration sampling time (AUClast) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.
Maximum observed concentration (Cmax) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.
Time to reach maximum observed concentration (Tmax) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.
Elimination half-life (T1/2) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.
Total body clearance (CL/F) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.
Apparent volume of distribution (V/F) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.
Area under the concentration-time curve from time zero to infinity (AUCinf) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.
Area under the concentration-time curve (AUC0-t) | Day 8
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as combination therapy.

CONTACTS AND LOCATIONS:
Locations (6):
- Novartis Investigative Site, Nanoro, Burkina Faso
- Novartis Investigative Site, Abidjan, Côte d’Ivoire
- Novartis Investigative Site, Libreville, Gabon
- Novartis Investigative Site, Kintampo, Ghana
- Novartis Investigative Site, Ahero, Kenya
- Novartis Investigative Site, Tororo, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.